CLINICAL TRIAL: NCT01738451
Title: A Two-Part Study to Evaluate the Effect of Repeat Oral Dosing of GSK2118436 on Cardiac Repolarization in Subjects With V600 BRAF Mutation-Positive Tumors: An Open-label, Dose-escalating Safety Lead-in Study Followed by a Single-sequence, Placebo-controlled, Single-blind Study
Brief Title: A Study to Evaluate the Effect of Repeat Oral Dosing of GSK2118436 on Cardiac Repolarization in Subjects With V600 BRAF Mutation-Positive Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113773
Record Dates: First submitted 2012-11-15; First posted 2012-11-30 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: ECG intervals and morphology; BRAF-mutation positive tumor; Holter monitor; BRAF inhibitor; GSK2118436; safety; cancer; QTc; pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1(Cohort 1): GSK2118436 225 mg (Experimental): GSK2118436 (3 capsules of 75 mg) will be administered orally at the dose of 225 mg BID from Day 1 to 7 (and single dose on Day 8) under fasted conditions, either 1 hour before or 2 hours after a meal.
  Interventions: Drug: GSK2118436 75 mg
- Part 1(Cohort 2): GSK2118436 300 mg (Experimental): GSK2118436 (4 capsules of 75 mg) will be administered orally at the dose of 300 mg BID from Day 1 to 7 (and single dose on Day 8) under fasted conditions, either 1 hour before or 2 hours after a meal. If 225 mg BID is not tolerated in Part 1 /Cohort 1, then Part 1/Cohort 2 will not be initiated and 150 mg BID will be used in Part 2.
  Interventions: Drug: GSK2118436 75 mg
- Part 2: GSK2118436 300 mg (or highest tolerated dose) (Experimental): Subjects will receive a single dose of GSK2118436/placebo (4 capsules of 75 mg/highest tolerated dose) orally on the first 2 days of the study followed by 2 doses daily for 6 days and a single dose on the 9th day. There will be 1 day when a placebo will be given. All doses will be administered under fasted conditions, either 1 hour before or 2 hours after a meal.
  Interventions: Drug: GSK2118436 75 mg; Drug: Placebo

INTERVENTIONS:
Drug: GSK2118436 75 mg — Each capsule contains 75 mg of GSK2118436A as the mesylate salt, micronized particles as active equivalents.
Drug: Placebo — Matching placebo capsules will be administered in Part 2 of the study.
  Arms: Part 2: GSK2118436 300 mg (or highest tolerated dose)

SUMMARY:
This is a Phase I, multicenter, 2-part study with Part 1 designed as a safety lead-in and Part 2 designed to evaluate the effect of GSK2118436 on cardiac repolarization (corrected QT interval [QTc] duration) as compared with placebo in subjects with V600 BRAF mutation-positive tumors.

Each part of the study will consist of screening (14 days prior to the start of the study treatment), treatment and follow-up period (14 days).

In Part 1 in Cohort 1 six subjects will receive GSK2118436 225 mg twice a day (BID) on study days 1 to 7 and a single 225 milligram (mg) dose on morning of Day 8. Based on the safety data of subjects in Cohort 1 subjects will be enrolled in Cohort 2 and the dose of GSK2118436 will be escalated to 300 mg BID. If the 225 mg dose of GSK2118436 is not well tolerated in Cohort 1 (i.e., 2 or more dose-limiting toxicities [DLTs]), then Cohort 2 of Part 1 will not be initiated and a dose of 150 mg BID of GSK2118436 will be administered in Part 2 of the study. In Cohort 2 six subjects will receive GSK2118436 300 mg BID on Study Days 1 to 7 and a single 300 mg dose on the morning of Day 8. Based on the safety data of subjects in Cohort 2 subjects will be enrolled in Part 2. If the 300 mg BID dose level of GSK2118436 is not well tolerated, then the highest tolerated dose will be selected for Part 2 of the study.

In Part 1 of the study the decision to proceed to the next cohort or Part 2 of the study will be based on the safety data of at least 6 evaluable subjects (<=1 DLTs during the 14 days following the first dose of GSK2118436).

In Part 2 of the study eligible subjects will receive a single dose of GSK2118436/placebo (4 capsules of 75 mg/highest tolerated dose) orally on the first 2 days of the study followed by 2 doses daily for 6 days and a single dose on the 9th day. There will be 1 day when a placebo will be given.

In both the parts of the study serial blood samples for pharmacokinetic (PK) analysis for GSK2118436 and its metabolites (GSK2285403, GSK2298683 and GSK2167542) will be obtained at the same time points on the first and last day of dosing (2nd day of dosing also included for Part 2). Safety electrocardiogram (ECG)s will be performed at several timepoints during the study. In Part 2 Holter ECG monitoring will be performed for 24 hours on the 1st, 2nd and 9th days of dosing.

ELIGIBILITY:
Inclusion Criteria:

* Has provided signed, written informed consent for this study.
* Male or female, age >=18 years of age at the time of signing the informed consent form
* Has confirmed diagnosis of a V600 BRAF-mutation positive tumor as determined by appropriate genetic testing.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has adequate baseline organ function as defined by: Absolute neutrophil count>=1.2 × 10^9/liter (L), hemoglobin>=9 gram (g)/deciliter (dL), platelets>= 75 × 10^9/L, prothrombin time (PT), international normalization ratio (INR) and partial thromboplastin time (PTT)<=1.3 times upper limit of normal (ULN), total bilirubin<=1.5 times ULN, alanine aminotransferase (ALT)<=2.5 times ULN; <5 times ULN if liver metastases are present, creatinine or<=1.5 times ULN, calculated creatinine clearance or 24-hour urine creatinine clearance>=60 mL/min and left ventricular ejection fraction (LVEF)>= institutional lower limit of normal (LLN) by echocardiogram (ECHO).
* For Part 2 subjects only: Have serum potassium, serum magnesium, and total serum calcium levels within normal limits.
* Able to swallow and retain orally administered medication and does not have any clinically significant GI abnormalities that may alter the absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* If a female subject of childbearing potential, must have a negative serum pregnancy test within 14 days of first dose of study treatment and agree to use effective contraception, during the study and for 4 weeks following the last dose of study treatment.

Exclusion Criteria:

* Known immediate or delayed hypersensitivity reaction to dabrafenib or excipients;
* Any of the following ECG findings: QT duration corrected using Fridericia's formula (QTcF) interval >450 milliseconds (msec), PR interval >220 msec or <=110 msec, bradycardia defined as sinus rate <50 beats per minute (bpm)
* Cardiac conduction abnormalities denoted by any of the following: evidence of second-degree (type II) or third-degree atrioventricular block, evidence of ventricular pre-excitation, electrocardiographic evidence of complete left bundle branch block (LBBB), intraventricular conduction delay with QRS duration >120 msec, evidence of atrial fibrillation or history of atrial fibrillation within the past 6 months or presence of cardiac pacemaker
* History of any one of the following cardiovascular conditions within the past 6 months: Class II, III, IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina or symptomatic peripheral vascular disease or other clinically significant cardiac disease
* LVEF, as measured by ECHO, below the institutional LLN, or if a LLN does not exist at an institution, <50%.
* Abnormal cardiac valve morphology (>=grade 2) documented by echocardiogram (subjects with minimal abnormalities [ie, mild regurgitation/stenosis] can be entered)
* Moderate valvular thickening
* Personal or immediate family history of long-QT syndrome.
* Anti-cancer therapy (e.g., chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or major surgery) within 21 days prior to enrolment; chemotherapy regimens without delayed toxicity within 14 days prior to enrollment; or use of an investigational anti-cancer drug within 28 days preceding the first dose of study treatment.
* Current use of a prohibited medication(s) or requires any of these medications during treatment with study treatment
* Current use of therapeutic warfarin.
* Unresolved toxicity of Grade 2 or higher from previous anticancer therapy, except alopecia or hemoglobin.
* A history of known Human Immunodeficiency Virus, Hepatitis B Virus (HBV), or Hepatitis C Virus infection. Subjects with documented laboratory evidence of HBV clearance may be enrolled.
* A history of known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Brain metastases that are: symptomatic, or treated (surgery, radiation therapy) but not clinically and radiographically stable 1 month after local therapy, or asymptomatic and untreated but >1 centimeter (cm) in the longest dimension
* Uncontrolled medical conditions (i.e., diabetes mellitus, hypertension), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol.
* History of another malignancy; Only (a) Subjects who have been successfully treated and are disease-free for 3 years, (b) a history of completely resected non-melanoma skin cancer, (c) successfully treated in situ carcinoma, (d) CLL in stable remission, or (e) indolent prostate cancer (definition: clinical stage T1 or T2a, Gleason score <=6, and PSA < 10 nanogram (ng)/mL) requiring no or only anti-hormonal therapy with histologically confirmed tumour lesions that can be clearly differentiated from lung cancer target and non-target lesions are eligible
* Pregnant or lactating/actively breastfeeding female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01-22 (Actual); Primary Completion 2014-11-28 (Actual); Study Completion 2014-11-28 (Actual)

PRIMARY OUTCOMES:
Part 1: Safety and tolerability of GSK2118436 as assessed by changes in physical examination findings | Screening, Day 1 and Week 6.
  Safety and tolerability parameter will include a complete (head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen [liver and spleen], lymph nodes, extremities, height and weight) and brief (skin, lungs, cardiovascular system, abdomen [liver and spleen] and weight) physical examination at Baseline and at the end of Part 1 of the study.
Part 1: Safety and tolerability of GSK2118436 as assessed by changes in vital signs measurements | Screening, pre-dose and 8 hours post-dose on Study Day 1, 8, 15, and Week 6.
  Safety and tolerability parameter will include measurement of vital signs (recording of systolic and diastolic blood pressure, temperature, and pulse rate) at Baseline and at the end of Part 1 of the study.
Part 1: Safety and tolerability of GSK2118436 as assessed by changes in ECG readings | Screening, Day 1, 8 Day 15 and Week 6. On study days 1 and 8, ECG will be obtained at 30 minutes pre-dose and 2-hours (hrs) post-dose administration.
  Safety and tolerability parameter will include ECGs readings (heart rate and measurement of RR, PR, QRS, QT, and QTc intervals) at Baseline and at the end of Part 1 of the study.
Part 1: Safety and tolerability of GSK2118436 as assessed by changes in clinical laboratory assessments | Day 1, 8, 15 and and Week 6.
  Safety and tolerability parameter will include laboratory values (hematology, clinical chemistry, coagulation, liver function tests, cardiac enzyme and beta-hCG/serum or urine pregnancy test for female subjects of childbearing potential only) at Baseline and at end of Part 1 of the study.
Part 2: Change from Baseline in QTcF interval at each time point for GSK2118436 | Baseline (Study Day -1)/pre-dose (Study Days 1 and 8) (within 30 minutes prior to administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, 10 and 24-hrs post-dose. Day 2 and 9, 24 hr post dose Holter ECG.
  Change from Baseline in QTcF interval at each time point for GSK2118436 will be calculated as average of 3 Holter ECG replicates per time point minus the value at Baseline.

SECONDARY OUTCOMES:
Part 1: Plasma concentration of GSK2118436 and its metabolites | On Day 1 and Day 8 at pre-dose (30 minutes (mins) prior to the administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, and 10-hours post-dose.
  Plasma concentrations of GSK2118436 and its metabolites GSK2285403, GSK2298683 and GSK2167542 will be recorded.
Part 1: The AUC(0-t)) of GSK2118436 and its metabolites | On Day 1 and Day 8 at pre-dose (30 mins prior to the administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, and 10-hours post-dose.
  Pharmacokinetic data will include area under the time-concentration curve from time zero (pre-dose) to last time of quantifiable concentration (AUC(0-t)) of GSK2118436 and its metabolites GSK2285403, GSK2298683 and GSK2167542.
Part 1: The Cmax of GSK2118436 and its metabolites | Part 1: Day 1 and Day 8 pre-dose (30 mins prior to the administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, and 10-hours post-dose.
  Pharmacokinetic data will include maximum plasma concentration (Cmax) of GSK2118436 and its metabolites GSK2285403, GSK2298683 and GSK2167542.
The Ctrough of GSK2118436 and its metabolites | Part 1: Day 8 pre-dose (30 mins prior to the administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, and 10-hours post-dose.
  Pharmacokinetic data will include predose concentration (Ctrough) of GSK2118436 and its metabolites GSK2285403, GSK2298683 and GSK2167542.
The tmax of GSK2118436 and its metabolites | Part 1: Day 1 and Day 8 pre-dose (30 mins prior to the administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, and 10-hours post-dose.
  Pharmacokinetic data will include time of occurrence of Cmax (tmax) of GSK2118436 and its metabolites GSK2285403, GSK2298683 and GSK2167542.
Part 2: Change from Baseline in slope of the relationships between the baseline-adjusted, placebo-corrected change in QTc interval and the plasma concentrations of GSK2118436 or its metabolites and predicted change in QTc | Part 2: Baseline (pre-dose study Days 1 and 8 within 30 minutes prior to administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, 10 and 24-hrs post-dose (Day 1 and 8). On Day 2 and 9, 24-hr post-dose PK sample and Holter ECG.
  The relationship between plasma concentrations of GSK2118436 and its metabolites (GSK2285403, GSK2298683 and GSK2167542) and the baseline-adjusted, placebo-corrected, time-matched change from Baseline in QTc intervals will be assessed.
Part 2: ECG parameters: and morphology assessments | Part 2: Baseline (pre-dose study Days 1 and 8 within 30 minutes prior to administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, 10 and 24-hrs post-dose (Day 1 and 8). On Day 2 and 9, 24-hr post dose Holter ECG.
  ECG parameters: QT, QTcB, QTci, HR, RR interval, PR interval, QRS interval and morphology will be assessed in subjects receiving GSK2118436.
Part 2: Plasma concentrations of GSK2118436 and its metabolites | On Days -1, 1 and 8 at pre-dose (within 30 minutes prior to administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hrs post-dose (Day 1 and 8). On Days 2 and 9 at 24-hr post dose PK sample.
  The plasma concentration of GSK2118436 and its metabolites GSK2285403, GSK2298683 and GSK2167542 will be measured.
The AUC(0-10) and AUC(0 t) of GSK2118436 and its metabolites (GSK2285403, GSK2298683 and GSK2167542) | Part 2: Days -1, 1 and 8: pre-dose (within 30 minutes prior to administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hrs post-dose (Day 1 and 8). On Day 2 and 9, 24-hr post dose PK sample.
  Pharmacokinetic data will include AUC from time zero (pre-dose) to 10 hours after the last dose of study treatment (AUC(0-10)) and AUC(0 t) of GSK2118436 and its metabolites GSK2285403, GSK2298683 and GSK2167542.
The AUC(0-infinity) of GSK2118436 and its metabolites (GSK2285403, GSK2298683 and GSK2167542) | Part 2: Day 1: pre-dose (within 30 minutes prior to administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hrs post-dose (Day 1).
  Pharmacokinetic data will include AUC from time zero to infinity AUC(0-infinity) of GSK2118436 and its metabolites GSK2285403, GSK2298683 and GSK2167542 on Study Day 1, if data permit).
The t½ of GSK2167542 and its metabolites | Part 2: Study Day 1 pre-dose (within 30 minutes prior to administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hrs post-dose.
  Pharmacokinetic data will include elimination half life (t1/2) of GSK2118436 and its metabolites GSK2285403, GSK2298683 and GSK2167542 if data permits.
Part 2: The Ctrough of GSK2167542 and its metabolites | Part 2: Study Day 8 pre-dose (within 30 minutes prior to administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hrs post-dose.
  Pharmacokinetic data will include C trough of GSK2118436 and its metabolites GSK2285403, GSK2298683 and GSK2167542.
Part 2: The Cmax, of GSK2167542 and its metabolites | Days -1, 1 and 8: pre-dose (within 30 minutes prior to administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hrs post-dose (Day 1 and 8). On Day 2 and 9, 24-hr post dose PK sample.
  Pharmacokinetic data will include Cmax of GSK2118436 and its metabolites GSK2285403, GSK2298683 and GSK2167542.
Part 2: The tmax, of GSK2167542 and its metabolites | Days -1, 1 and 8: pre-dose (within 30 minutes prior to administration of study treatment) and 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hrs post-dose (Day 1 and 8). On Day 2 and 9, 24-hr post dose PK sample.
  Pharmacokinetic data will include tmax of GSK2118436 and its metabolites GSK2285403, GSK2298683 and GSK2167542.
Part 2: Safety of GSK2118436 as assessed by number of subjects with adverse events (AE)s | Continuous throughout the study.
  Safety parameters will include recording of AEs, in Part 2 of the study.
Part 2: Safety of GSK2118436 as assessed by changes in vital signs measurements | Screening, Day -1, Day 1, Day 8, Day 9 and Week 5.
  Safety parameters will include measurement of vital signs (recording of systolic and diastolic blood pressure, temperature, and pulse rate) at Baseline and at the end of Part 2 of the study.
Part 2: Safety of GSK2118436 as assessed by changes in ECG readings | Screening, Day -1, Day 1, Day 2, Day 8, Day 9 and Week 5.
  Safety parameters will include ECGs readings (heart rate and measurement of RR, PR, QRS, QT, and QTc intervals) at Baseline and at the end of Part 2 of the study.
Part 2: Safety of GSK2118436 as assessed by changes in clinical laboratory assessments | Screening, Day -1, Day 1, Day 8, Day 9 and Week 5.
  Safety parameters will include laboratory values (hematology, clinical chemistry, coagulation, liver function tests, cardiac enzyme and beta-hCG/serum or urine pregnancy test for female subjects of childbearing potential only) at Baseline and at end of Part 2 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (5):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
- Australia (2):
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Nebot N, Arkenau HT, Infante JR, Chandler JC, Weickhardt A, Lickliter JD, Sarantopoulos J, Gordon MS, Mak G, St-Pierre A, Tang L, Mookerjee B, Carson SW, Hayes S, Grossmann KF. Evaluation of the effect of dabrafenib and metabolites on QTc interval in patients with BRAF V600-mutant tumours. Br J Clin Pharmacol. 2018 Apr;84(4):764-775. doi: 10.1111/bcp.13488. Epub 2018 Jan 23. PMID 29243287
- See also: Results for study 113773 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113773?search=study&search_terms=113773#rs